CLINICAL TRIAL: NCT02814045
Title: Impact of Obstructive Sleep Apnea in the Evolution of Alzheimer Disease. Role of Hypoxia and Sleep Fragmentation
Brief Title: Role of Hypoxia Ans Sleep Fragmentation in Alzheimer's Disease. and Sleep Fragmentation.
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, PhD, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: 464/C/2014
Record Dates: First submitted 2015-12-05; First posted 2016-06-27 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer's Disease; Obstructive Sleep Apnea
Keywords: biomarkers, sleep fragmentation, intermittent hypoxia
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea, Obstructive; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — APoE4
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alzheimer with OSA: Alzheimer with OSA after PSG
- Alzheimer without OSA: Alzheimer without OSA after PSG

SUMMARY:
Alzheimer's Disease (AD) is the most prevalent neurodegenerative disease, manifested as an initial deficit of episodic memory that evolves into a global cognitive and psychosocial dysfunction and which prevalence is increasing around the world. Sleep disturbance is frequent since early stages of the disease and sleep fragmentation had been demonstrated increase the production of amyloid peptide (AB) (main pathological hallmark) in non-demented population. Obstructive Sleep Apnea (OSA), which consist in intermittent hypoxia and sleep fragmentation, is a major health problem with multiple systemic effects and it's very prevalent in AD. However, the influence of this comorbidity on the cognitive evolution of AD patients remains unknown. The investigation of neurobiological markers and sleep recording may reveal potential mechanisms of neurodegeneration and explain the influence of sleep fragmentation and/or hypoxia on cognitive decline.

To fill those gaps, investigators will perform a multidisciplinary and translational project to assess the progression of symptoms in AD patients, diagnosis of sleep disturbance and new biomarkers of progression of the disease.

The present proposal is going to be developed by coordination of different expertises that will be range from the clinical research conducted by a medical neurologist, to the animal model and most molecular work, to be done by an experimented group in mouse work.

DETAILED DESCRIPTION:
As AD and OSA have a bidirectional relationship, OSA causes cerebral hypoxia and sleep fragmentation favouring the deposition of AB and AD causes alterations in sleep quality, investigators will develop a comprehensive project with human patients and an animal model of AD with sleep fragmentation (SF) and intermittent hypoxia (IH).

Investigators prospectively will study consecutive patients with new diagnosis of mild probable Alzheimer's Disease by a neurologist. Investigators will define Alzheimer's Disease according to National Institute of Aging-Alzheimer's Association criteria (NIA-AA).

All patients undergo routine neuropsychological battery, sleep polysomnography and actigraphy registry, brain MRI, lumbar puncture and blood biochemistry.

Neuropsychological battery The following assessments will be used at baseline and at 12 months: Alzheimer's Disease Assessment Scale-cognitive (ADAS-cog), Mini-Mental State Exam (MMSE), Hachinski Scale, Digit Wechsler Adult Intelligence Scale(WAIS- III); Stroop Color-Word Interference Test (Stroop); Verbal fluency test; Trail Making Test (TMT) A and B; California verbal learning test (CVLT), Rey-Osterrieth Complex Figure Test (RCFT), Cornell depression scale, neuropsychiatric inventory, caregiver burden scale and EuroQol Test.

CSF Cerebrospinal fluid will be obtained by lumbar punction at 8 am, after overnight fasting. Amyloid beta 42 (AB42), tau and phosphotau will be measured using enzyme-linked immunoabsorbent assay (ELISA)(INNOTEST, Innogenetics). The cut-off will be based on prior studies of our laboratory. Also, ELISA will be employed to detect the levels of hypoxia-inducible factor 1-alpha (HIF-1alpha vascular endothelial growth factor (VEGF), nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF) in the cerebrospinal fluid (CSF).

Sleep measurement To evaluate the sleep characteristics of patients a PSG will be done to all patients at baseline. The duration of each PSG will be about 8 hours, from about 23 pm until 7 pm. 6 channels of EEG will be recorded with reference to the two ears.

Channels included 2 central electroencephalograms (EEG), bilateral electrooculogram (EOG), chin electromyogram (EMG), thoracic and abdominal respiratory effort, airflow (using nasal-oral thermocouple and nasal pressure recording), finger pulse oximetry, electrocardiogram (ECG), body position, and bilateral piezoelectric sensors to detect leg movements. Data will be evaluated by trained technicians, and sleep stage will be assessed in 30-second epochs according to standard criteria. Apnea (complete cessation of airflow) and hypopnea (discernible > 30% reduction in airflow) will be defined if occurring for 10 seconds or longer and accompanied by a 4% or greater oxygen desaturation. Arousals from sleep will be defined as an abrupt shift in EEG frequency of 3 seconds or longer; arousals during rapid eye movement (REM) sleep required an increase in chin EMG activity. Sleep disordered breathing will be measured by the apnea-hypopnea index (AHI; the number of apnea plus hypopnea events per hour of sleep), and prevalent sleep-disordered breathing coded as the apnea -hypopnea index of 15 or more events per hour. Calculated variables used as indices of hypoxia included the oxygen 4%15 or < 15 events per hour; the percentage of sleep time with oxygen saturation (SaO2) < 90% 1% of sleep time or < 1% sleep time with SaO2 < 90%; and the percentage of sleep time in apnea or hypopnea (>4% of oxygen desaturation coded into tertiles). Calculated variables of sleep fragmentation will include arousal index (AI) defined as the number of arousals per hour of sleep and minutes of wake after sleep onset (WASO) (both coded into tertiles). Sleep duration will be measured as the total sleep time (TST) coded into tertile. Investigators also measured REM and stage I sleep duration.Patterns of sleep and circadian rhythms will be measured with an actigraph (Actiwatch 2; Philips). Participants will be instructed to wear an actigraph on the nondominant wrist for 14 days and to push a marker on the actigraph whenever getting in and out of bed. The quantity of sleep will be measured with total sleep time. The quality of sleep will be measured with sleep efficiency, which is total sleep time divided by time in bed, expressed as a percentage. A secondary measure of sleep quality will be wake time after sleep onset. Concurrently, participants filled out a sleep diary each morning. The sleep diary queried for naps the previous day, bedtime, sleep latency, nighttime awakenings, wake time, and opened comment. The number of days per week that at least 1 nap will be taken was calculated as "nap days per week." Brain MRI

All patients will be evaluated by MRI performed using a Siemens Avant 1.5 T, MRI scanner. The protocol performed will include:

1. Volumetric T1-weighted 3D multiplanar reconstruction, FoV 256 mm, slice thickness 1 mm, Time relapse (TR) 1600 ms, TE 3,01 ms, distance factor 50%. T2 tse axial, FoV 230 mm, slice thickness 5 mm, TR 3560 ms, TE 89 ms, distance factor 30%. Flair axial, FoV 230 mm, slice thickness 5 mm, TR 8000 ms, Time exposition (TE) 94 ms, distance factor 30%. T2 gradient echo axial, FoV 230 mm, slice thickness 5 mm, TR 800 ms, TE 26 ms, distance factor 30%. Echoplanar diffusion images, FoV 230 mm, slice thickness 5 mm, Time relapse 3902 ms, TE 102 ms, distance factor 40%. T2 Turbo spin echo coronal, FoV 210 mm, slice thickness 5 mm, TR 3250 ms, TE 100 ms, distance factor 20%.
2. Perfusion - weighted images (PWI) will be obtained using an echo-planar imaging sequence (FoV 230 mm, slice thickness 5 mm, TR 1439 ms, TE 30 ms) after the injection of a gadolinium chelate (Gadovist) using an automatic injector with a flow of 4 ml/s.
3. Spectroscopy Study evaluating the cortical gray matter of the posterior cingulate and right middle temporal gyrus with the use of two echo times (31 and 136 ms) and the same TR 2000 ms. Dimensions of the volume in posterior cingulate 20 x 20 x 20 mm (8 cc) and right middle temporal gyrus 18 x 18 x 18 mm (5,8 cc). The posterior cingulate will be taken as the reference due to it is the most affected region in patients with Alzheimer in SPECT studies.

Metabolomic and lipidaemic analyses. Lipidaemic and metabolomic analyses will be performed on the blood sample and CSF. For metabolites extraction, samples will be deproteinized using cold methanol in the presence of antioxidants and internal standards. Lipids will be extracted using chloroform/methanol in the presence of antioxidants and class-specific internal standards. Metabolite and lipid extracts will be subjected to mass spectrometry using an High pressure liquid chromatography 1290 series coupled to an Electrospray ionization-quadrupole reflection time-of-flight (ESI-QTOF) Mass spectrometry/Mass Spectrometry 6520 (Agilent Technologies, Santa Clara, California, USA). The liquid chromatography-mass spectrometry metabolomic and lipidemic analyses will be based on previously described methods (Jove et al., 2013; Jove et al., 2014).

Blood samples Blood samples will be obtained by a venous puncture at 8 am after PSG. The samples will be processed and stored in accordance with Royal Decree 1716/2011 of 18th November 2011 by authorization requirements and operation of biobanks for biomedical research and treatment of biological samples down of human origin (BOE No. 290 of 12.12.2011).

Determination of molecular markers, metabolomics, lipidemic will be drawn. Commercial biomarkers (TNF-alpha, Interleukine-6 and Interleukine-8), the Thiobarbituric Acid Reactive Substances (TBARS) will be measured. Will be performed genotyping APOE4.

Sample size calculation This is an observational cohort study, which will include a group of 72 patients with OSA and another 72 patients without OSA from the same population of patients with mild initial AD after making PSG. Patients will be recruited consecutively. If more patients with AD that the ability to carry out the study of sleep, investigators will apply a random selection (web based tool).

The sample size has been calculated accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast to detect a difference equal to or greater than 3.5 units on the ADAS-cog scale. It is assumed that the common standard deviation is 7. It has been estimated a loss rate of 12% follow-up.

Statistical analysis The standard statistical analysis will be performed with the SPSS statistical package, version 15.0 (SPSS, Chicago, Illinois,USA). The results of the different variables will be expressed as means ± standard deviation value. The statistical significance of differences between groups and variables assessed by analysis of variance (ANOVA) considering the practice of repeated measurements of the same variable. To investigate the existence of correlations between clinical variables will use in bivariate Spearman correlation test and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed of mild probable AD according to NIA-AA criteria (MMSE>20).
2. Informed Consent Form signed by the patient (and/or if applicable the legal representative if different from the responsible caregiver) and the responsible caregiver.
3. The patient has a knowledgeable and reliable caregiver who will accompany the patient to all clinic visits during the study.
4. Absence of visual and hearing problems that, in the investigator's judgement, difficult for compliance with the study procedures.

Exclusion Criteria:

1. Previous diagnosis of OSA.
2. Severe Alzheimer's disease, other types of dementia or patients with mild Alzheimer's disease with current acetylcholinesterase inhibitors or memantine treatment.
3. Presence of any previously diagnosed sleep disorder: narcolepsy, insomnia, chronic lack of sleep.
4. Having serious comorbidities: cancer, excessive intake of alcohol (>280 gr/week), severe depression, severe renal or hepatic insufficiency, severe cardiac or respiratory failure.
5. Currently receiving an investigational drug or device.
6. Patient or family declining to take part.
7. Disabling drowsiness not justifiable by any other cause.
8. The patient has MRI evidence of hydrocephalus, stroke, a space-occupying lesion, cerebral infection or any clinically significant central nervous system disease other than AD.
9. The patient suffers from mental retardation, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
10. The patient has an untreated vitamin B12 or folate deficiency that is considered clinically significant, or has clinical and laboratory evidence of untreated thyroid disease. Patients with vitamin B12 or folate deficiency may be enrolled in the study provided they have been on a supplement therapy for >3 months prior to the Screening Visit and are stable. Patients with thyroid disease may be enrolled in the study provided they are stable and euthyroid.
11. Patient on betablockers, antidepressants, neuroleptics, hypnotics, or they have been removed 15 days before conducting polysomnography (PSG).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We prospectively will studied consecutive patients with new diagnosis of mild probable Alzheimer's Disease by a neurologist. We will define Alzheimer's Disease according NIA-AA criteria.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive scores on the Disease Assessment Scale-cognitive at 12 months in patients with mild AD with and without OSA. | One year
  For this objective we will recruit consecutively 72 patients with OSA and another 72 patients without OSA from the same population of patients with mild initial AD. We will use extensive neuropsychological battery at baseline and at 12 month and polysomnography (PSG) to select both groups of patients at baseline.

SECONDARY OUTCOMES:
Differential pattern of biomarkers at baseline in in patients with mild AD with and without OSA. | One year
  For this objective we will use CSF (ELISA will be employed to detect the levels of hypoxia-inducible factor 1-alpha (HIF-1alpha), vascular endothelial growth factor (VEGF), nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF); and CSF biomarkers of AD as AB42, tau and phosphotau. Lipidaemic and metabolomic analyses will be performed on both, blood sample and CSF. Brain MRI (hippocampal volume, specific patterns of cerebral perfusion and spectroscopy) and actigraph registry. Blood samples to determine inflammatory markers (TNF-alpha, Interleukine-6 and Interleukine-8), the Thiobarbituric Acid Reactive Substances (TBARS) and genotyping APOE4 will be preformed. We will analyze the correlation of these biological biomarkers with cognitive and behavioural progression in OSA and non-OSA AD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Piñol, Md;PhD, Principal Investigator — Hospital Santa Maria
Locations (2):
- Spain (2):
  - Hospital santa Maria, Lleida, Catalonia
  - Hospital Santa Maria Lleida, Lleida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dakterzada F, Benitez ID, Targa A, Carnes A, Pujol M, Jove M, Minguez O, Vaca R, Sanchez-de-la-Torre M, Barbe F, Pamplona R, Pinol-Ripoll G. Blood-based lipidomic signature of severe obstructive sleep apnoea in Alzheimer's disease. Alzheimers Res Ther. 2022 Nov 3;14(1):163. doi: 10.1186/s13195-022-01102-8. PMID 36329512
- [Derived] Targa ADS, Benitez ID, Dakterzada F, Carnes A, Pujol M, Jorge C, Minguez O, Dalmases M, Sanchez-de-la-Torre M, Barbe F, Pinol-Ripoll G. Sleep profile predicts the cognitive decline of mild-moderate Alzheimer's disease patients. Sleep. 2021 Oct 11;44(10):zsab117. doi: 10.1093/sleep/zsab117. PMID 33969423
- [Derived] Jorge C, Targa A, Benitez ID, Dakterzada F, Torres G, Minguez O, Carnes A, Pujol M, Gibert A, Lopez R, Gaeta AM, Dalmases M, Farre R, Sanchez-de-la-Torre M, Barbe F, Pinol-Ripoll G. Obstructive sleep apnoea and cognitive decline in mild-to-moderate Alzheimer's disease. Eur Respir J. 2020 Nov 19;56(5):2000523. doi: 10.1183/13993003.00523-2020. Print 2020 Nov. PMID 32554539